CLINICAL TRIAL: NCT01751126
Title: A Multicenter, Randomized, Double-Masked, 3 Parallel Arms, Placebo Controlled Study to Assess the Efficacy and Safety of NOVA22007 1mg/mL (Ciclosporin/Cyclosporine) Eye Drops, Emulsion Administered in Paediatric Patients With Active Severe Vernal Keratoconjunctivitis With Severe Keratitis
Brief Title: Double-Masked Trial of NOVA22007 (1mg/mL Ciclosporin/Cyclosporine) Versus Vehicle in Pediatric Patients With Active Severe Vernal Keratoconjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NVG09B113
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Results first posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Vernal Keratoconjunctivitis
Keywords: vernal keratoconjunctivitis; ciclosporin; cyclosporine
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ciclosporin (Experimental): One drop of ciclosporin (NOVA22007) 1 mg/ml 4 times a day as monotherapy (morning, noon, afternoon and evening).
  Interventions: Drug: NOVA22007 ''Ciclosporin''
- Ciclosporin/Placebo (Experimental): One drop of ciclosporin (NOVA22007) 1 mg/ml twice a day and one drop of placebo twice a day (active study treatment morning and evening and placebo noon and afternoon) as monotherapy.
  Interventions: Drug: NOVA22007 ''Ciclosporin''; Drug: Placebo
- Placebo (Placebo Comparator): One drop of placebo 4 times a day as monotherapy (morning, noon, afternoon and evening).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NOVA22007 ''Ciclosporin'' — Sterile, ophthalmic cationic oil-in-water emulsion containing 1 mg/ml Ciclosporin.
  Arms: Ciclosporin; Ciclosporin/Placebo
Drug: Placebo — Sterile, drug-free, cationic ophthalmic oil-in-water emulsion containing 0 mg/ml Ciclosporin.
  Arms: Ciclosporin/Placebo; Placebo

SUMMARY:
The objective of this study is to compare the efficacy of two different dosing regimen of NOVA22007 (1mg/ml ciclosporin/cyclosporine) eye drops, emulsion versus placebo (vehicle of the formulation) administered four times a day in patients with severe vernal keratoconjunctivitis after 4 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males or females from 4 to less than 18 years of age.
* History of at least one recurrence of vernal keratoconjunctivitis (VKC) in the past year prior to enrolment.
* Patients not receiving any treatment for an established and active VKC; or patients already receiving treatment for their VKC provided treatment is stopped according to the wash-out period specified in the exclusion criteria.
* Active severe VKC consistent with grade 3 or 4 of Bonini scale (Bonini 2007) with severe keratitis (grade 4 or 5 on the modified Oxford scale).
* Mean score of 4 subjective symptoms (photophobia, tearing, itching and mucous discharge) ≥ 60 mm using a 100 mm Visual Analogue Scale (where "0" means no symptom and "100" means the worst that have been ever experienced).

Exclusion Criteria:

* Any relevant ocular anomaly other than VKC interfering with the ocular surface including trauma, post radiation keratitis, severe blepharitis, rosacea, corneal ulcer etc.
* Abnormal lid anatomy, abnormalities of the nasolacrimal drainage system or blinking function in either eye.
* Active herpes keratitis or history of ocular herpes.
* Active ocular infection (viral, bacterial, fungal, protozoal).
* Any ocular diseases other than VKC requiring topical ocular treatment during the course of the study.
* Contact lenses wear during the study.
* Topical and/or systemic use of corticosteroids within one week prior to enrolment.
* Topical ciclosporin (e.g. Restasis®), tacrolimus or sirolimus within 90 days prior to enrolment.
* Scraping of the vernal plaque within one month prior to the Baseline visit.
* Ocular surgery within 6 months prior to the Baseline visit (excluding surgical treatment of the vernal plaque).
* Disease not stabilized within 30 days before the Baseline Visit (e.g., diabetes with glycemia out of range, thyroid malfunction, uncontrolled autoimmune disease, current systemic infections) or judged by the investigator to be incompatible with the study.
* Presence or history of severe systemic allergy.
* Any systemic immunosuppressant drugs within 90 days before the Baseline Visit.
* Known hypersensitivity to one of the components of the study or procedural medications (e.g., fluorescein, etc).
* History of malignancy in the last 5 years.
* Pregnancy or lactation at the Baseline Visit.
* History of ocular varicella-zoster or vaccinia virus infection.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 169 (Actual)
Dates: Start 2013-04-29; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (4):
  - Glendale, CA, USA, Glendale, California
  - Irvine, CA, USA, Irvine, California
  - Rancho Cordova, CA, USA, Rancho Cordova, California
  - Miami, FL, USA, Miami, Florida
- Zagreb, City of Zagreb, HR, Zagreb, City of Zagreb, Croatia
- France (5):
  - Marseille, Bouches-du-Rhône, FR, Marseille, Bouches-du-Rhône
  - Angers CEDEX 9, Maine-et-Loire, FR, Angers, Maine-et-Loire
  - Amiens CEDEX, Somme, FR, Amiens, Somme
  - Tours CEDEX 9, FR, Tours
  - Paris CEDEX 8, Île-de-France, FR, Paris, Île-de-France Region
- Mainz, Rhineland-Palatinate, DE, Mainz, Rhineland-Palatinate, Germany
- Greece (3):
  - Ioannina, Eprius, GR, Ioannina, Eprius
  - Thessaloniki, Macedonia, GR, Thessaloniki, Macedonia
  - Larissa, Thessaly, GR, Larissa, Thessaly
- Hungary (3):
  - Szeged, Csongrád, HU, Szeged, Csongrád megye
  - Debrecen, Hajdú-Bihar, HU, Debrecen, Hajdú-Bihar
  - Budapest, HU, Budapest
- India (4):
  - Visakhapatnam, Andhra Pradesh, IN, Visakhapatnam, Andhra Pradesh
  - New Delhi, National Capitol Territory, IN, New Delhi, National Capitol Territory
  - Chennai, Tamil Nadu, IN, Chennai, Tamil Nadu
  - Lucknow, Uttar Pradesh, IN, Lucknow, Uttar Pradesh
- Israel (5):
  - Be'er-Sheva, IL, Beersheba
  - Jerusalem, IL, Jerusalem
  - Petah-Tikva, IL, Petah Tikva
  - Rehovot, IL, Rehovot
  - Tel-Aviv, IL, Tel Aviv
- Italy (6):
  - Bologna, Emilia-Romagna, IT, Bologna, Emilia-Romagna
  - Lavagna, Liguria, IT, Lavagna, Liguria
  - Cinisello, Pisa, IT, Cinisello Balsamo, Pisa
  - Firenze, Tuscany, IT, Florence, Tuscany
  - Padova, Veneto, IT, Padua, Veneto
  - Messina, Messina, IT, Messina
- Portugal (2):
  - Vila Nova de Gaia, Douro Litoral, PT, Vila Nova de Gaia, Douro Litoral
  - Lisboa, Extremadura, PT, Lisbon, Extremadura
- Spain (9):
  - Torrevieja, Alicante, ES, Torrevieja, Alicante
  - Barakaldo, Biscay, ES, Barakaldo, Biscay
  - San Sebastián, Guipúzcoa, ES, San Sebastián, Guipúzcoa
  - Aranjuez, Madrid, ES, Aranjuez, Madrid
  - A Coruña, A Coruña, ES, A Coruña
  - Alicante, Alicante, ES, Alicante
  - Madrid, Madrid, ES, Madrid
  - Sevilla, Sevilla, ES, Seville
  - Valencia, Valencia, ES, Valencia

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose Regimen: 1 drop of CsA (NOVA22007) 1 mg/mL 4 times a day as monotherapy (morning, noon, afternoon and evening).
- Low Dose Regimen: 1 drop of CsA (NOVA22007) 1 mg/mL twice a day and 1 drop of placebo twice a day (active study treatment morning and evening and placebo noon and afternoon) as monotherapy.
- Placebo: 1 drop of placebo 4 times a day as monotherapy.
Period: Period I
Arm/Group | High Dose Regimen | Low Dose Regimen | Placebo
Started | 57 | 54 | 58
Completed | 51 | 43 | 49
Not Completed | 6 | 11 | 9
Period: Period II
Arm/Group | High Dose Regimen | Low Dose Regimen | Placebo
Started | 72 | 70 | 0 (Following completion of the first period of the trial, all patients were to be administered NOVA22007 (High or Low dose) for a safety 8-month follow-up period.)
Completed | 72 | 70 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One participant from the High dose regimen withdrew at the first week of randomization and not related to study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Regimen | Low Dose Regimen | Placebo | Total
Number analyzed (Participants) | 56 | 54 | 58 | 168
Age, Customized [Mean (Standard Deviation); unit: years]
  Children (4-18 years) | 9.1 (3.3) | 9.6 (3.4) | 8.9 (3.2) | 9.2 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 12 | 36
  Male | 44 | 42 | 46 | 132
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 11 | 11 | 13 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 2 | 10
  White | 40 | 38 | 41 | 119
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Average Penalties Adjusted Composite Efficacy Score (CFS) Score Over the 4 Months
Description: Efficacy was assessed every month during the 4-month treatment phase and compared with Baseline using a composite criterion based on:
  * Keratitis assessed by the modified Oxford scale (7-point ordinal scale, score 0, 0.5, and 1 to 5). On this modified scale, the score 0 corresponded to no staining dots and the score 0.5 to three or less staining dots. A CFS grade of 0 represented complete corneal clearing.
  * Need for rescue medication.
  * Occurrence of corneal ulceration.
  An efficacy score was calculated as follows:
  Patient's score at month X = CFS (Baseline) - CFS (Month X) + penalty (ies) Penalty for rescue medication: -1 (per course, with a maximum of 2 courses between 2 scheduled visits) Penalty for corneal ulceration: -1 (per occurrence).
  A positive value indicated improvement.
  The maximum CFS is five and the minimum cannot be set due to the number of rescue medication and ulceration which decreases the penalty adjusted CFS.
Time Frame: over the 4 months
Measure: Mean (Standard Deviation); unit: Penalties Adjusted CFS Score
Arm/Group | High Dose Regimen | Low Dose Regimen | Placebo
Number analyzed (Participants) | 56 | 54 | 58
Penalties Adjusted CFS Score | 2.06 (1.44) | 1.93 (1.37) | 1.34 (1.22)
Statistical Analysis 1: Comparison: High Dose Regimen vs Placebo; Test type: Superiority; p = 0.007, t-test, 2 sided — ANCOVA with treatment as well as the baseline CFS and the exposure to Vernal keratoconjunctivitis (VKC) seasons (Hochberg procedure); LS Mean = 0.76, 95% CI 2-sided [0.26 to 1.27]
Statistical Analysis 2: Comparison: Low Dose Regimen vs Placebo; Test type: Superiority; p = 0.010, ANCOVA; ANCOVA with treatment as well as the baseline CFS and the exposure to Vernal keratoconjunctivitis (VKC) seasons (Hochberg procedure); LS Mean = 0.67, 95% CI 2-sided [0.16 to 1.18]

2. Secondary Outcome: Best Corrected Distance Visual Acuity (BCDVA) in 4-month Randomized Period I
Description: Best corrected distance visual acuity (BCDVA) was measured with the patient's best correction and recorded in LogMAR (log of the Minimum Angle of Resolution) A negative LogMar BCDVA measure shows an improvement, whereas positive values indicates poor vision.
Time Frame: Up to Month4
Population: SS population
Measure: Mean (Standard Deviation); unit: letters
Groups:
- LogMAR - High Dose Regimen: Logarithm of the Minimum Angle of Resolution (LogMAR)
Arm/Group | LogMAR - High Dose Regimen | LogMAR - Low Dose Regimen | LogMAR-Placebo | Change From Baseline in LogMAR- High Dose | Change From Baseline in LogMAR- Low Dose | Change From Baseline in LogMAR- Placebo
Number analyzed (Participants) | 57 | 54 | 58 | 57 | 54 | 58
letters
  Analysis Eye-Baseline: number analyzed (Participants) | 57 | 54 | 57 | 57 | 54 | 58
  Analysis Eye-Baseline | 0.293 (0.297) | 0.209 (0.284) | 0.302 (0.347) | 0 (0) | 0 (0) | 0 (0)
  Analysis Eye-Month 1: number analyzed (Participants) | 55 | 48 | 55 | 55 | 48 | 55
  Analysis Eye-Month 1 | 0.263 (0.292) | 0.160 (0.241) | 0.285 (0.362) | -0.036 (0.187) | -0.058 (0.199) | -0.027 (0.182)
  Analysis Eye-Month 2: number analyzed (Participants) | 54 | 46 | 51 | 54 | 46 | 51
  Analysis Eye-Month 2 | 0.221 (0.251) | 0.146 (0.214) | 0.331 (0.352) | -0.071 (0.191) | -0.073 (0.202) | 0.003 (0.233)
  Analysis Eye-Month 3: number analyzed (Participants) | 52 | 44 | 49 | 52 | 44 | 49
  Analysis Eye-Month 3 | 0.172 (0.235) | 0.110 (0.204) | 0.273 (0.318) | -0.110 (0.173) | -0.089 (0.233) | -0.066 (0.229)
  Analysis Eye-Month 4: number analyzed (Participants) | 51 | 43 | 48 | 51 | 43 | 48
  Analysis Eye-Month 4 | 0.149 (0.244) | 0.097 (0.203) | 0.237 (0.308) | -0.127 (0.165) | -0.110 (0.233) | -0.109 (0.211)
  Analysis Eye-Month 4/ Early Termination: number analyzed (Participants) | 56 | 51 | 55 | 56 | 51 | 55
  Analysis Eye-Month 4/ Early Termination | 0.158 (0.249) | 0.114 (0.212) | 0.217 (0.295) | -0.135 (0.220) | -0.091 (0.257) | -0.097 (0.210)

3. Secondary Outcome: Best Corrected Distance Visual Acuity (BCDVA) in 8-month Safety FU Period- Period II
Description: Best corrected distance visual acuity (BCDVA) was measured with the patient's best correction and recorded in LogMAR (log of the Minimum Angle of Resolution) A negative LogMar BCDVA measure shows an improvement, whereas positive values indicate poor vision.
Time Frame: Up to Month12
Population: SS population
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | LogMAR - High Dose Regimen | LogMAR - Placebo | LogMAR-Total | Change From Baseline in LogMAR- High Dose | Change From Baseline in LogMAR- Placebo | Change From Baseline in LogMAR- Total
Number analyzed (Participants) | 50 | 22 | 72 | 50 | 22 | 72
letters
  Analysis Eye-Baseline (Month 4): number analyzed (Participants) | 50 | 21 | 71 | 50 | 22 | 72
  Analysis Eye-Baseline (Month 4) | 0.152 (0.246) | 0.250 (0.317) | 0.181 (0.270) | 0 (0) | 0 (0) | 0 (0)
  Analysis Eye-Month 6: number analyzed (Participants) | 50 | 22 | 72 | 50 | 21 | 71
  Analysis Eye-Month 6 | 0.128 (0.230) | 0.258 (0.359) | 0.168 (0.280) | -0.024 (0.114) | -0.017 (0.143) | -0.022 (0.122)
  Analysis Eye-Month 8: number analyzed (Participants) | 49 | 21 | 70 | 49 | 21 | 70
  Analysis Eye-Month 8 | 0.141 (0.228) | 0.222 (0.324) | 0.165 (0.261) | -0.015 (0.136) | -0.029 (0.155) | -0.019 (0.141)
  Analysis Eye-Month 10: number analyzed (Participants) | 49 | 21 | 70 | 49 | 21 | 70
  Analysis Eye-Month 10 | 0.141 (0.222) | 0.207 (0.325) | 0.160 (0.257) | -0.014 (0.149) | -0.044 (0.128) | -0.023 (0.143)
  Analysis Eye-Month 12: number analyzed (Participants) | 49 | 21 | 70 | 49 | 21 | 70
  Analysis Eye-Month 12 | 0.134 (0.214) | 0.220 (0.363) | 0.160 (0.268) | -0.020 (0.152) | -0.030 (0.172) | -0.023 (0.157)
  Analysis Eye-Month 12/ Early Termination: number analyzed (Participants) | 50 | 21 | 71 | 50 | 21 | 71
  Analysis Eye-Month 12/ Early Termination | 0.136 (0.212) | 0.220 (0.363) | 0.161 (0.266) | -0.016 (0.154) | -0.030 (0.172) | -0.020 (0.158)

4. Secondary Outcome: Number of Courses of Rescue Medication in Period I
Description: Use of rescue medication: the total number of topical corticosteroid courses was assessed at each visit during the 4-month efficacy evaluation treatment period.
Time Frame: Up to Month4
Population: Participants reduced due to missing data
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Regimen | Low Dose Regimen | Placebo
Number analyzed (Participants) | 56 | 54 | 58
Participants
  Month1, zero course: number analyzed (Participants) | 54 | 50 | 57
  Month1, zero course | 51 | 41 | 44
  Month 1, one course: number analyzed (Participants) | 54 | 50 | 57
  Month 1, one course | 3 | 7 | 11
  Month1, two courses: number analyzed (Participants) | 54 | 50 | 57
  Month1, two courses | 0 | 2 | 2
  Month2, zero course: number analyzed (Participants) | 53 | 47 | 52
  Month2, zero course | 45 | 43 | 38
  Month 2, one course: number analyzed (Participants) | 53 | 47 | 52
  Month 2, one course | 6 | 2 | 11
  Month 2, two courses: number analyzed (Participants) | 53 | 47 | 52
  Month 2, two courses | 2 | 2 | 3
  Month3, zero course: number analyzed (Participants) | 51 | 46 | 50
  Month3, zero course | 43 | 42 | 34
  Month3, one course: number analyzed (Participants) | 51 | 46 | 50
  Month3, one course | 7 | 2 | 12
  Month 3, two courses: number analyzed (Participants) | 51 | 46 | 50
  Month 3, two courses | 1 | 2 | 4
  Month4, zero course: number analyzed (Participants) | 50 | 44 | 48
  Month4, zero course | 42 | 41 | 38
  Month4, one course: number analyzed (Participants) | 50 | 44 | 48
  Month4, one course | 6 | 2 | 8
  Month 4, two courses: number analyzed (Participants) | 50 | 44 | 48
  Month 4, two courses | 2 | 1 | 2
  Month 4/Early Termination, zero course | 46 | 46 | 43
  Month 4/Early Termination, one course | 7 | 5 | 11
  Month 4/Early Termination, two courses | 3 | 3 | 4

ADVERSE EVENTS:
Time Frame: From the time the informed consent form was signed until the last study visit at Month 12.
Groups:
- .1% QID (4 Months) Plus .1% QID (8 Months Safety Follow-up): Participants in this group received High dose in Period I (4 months) and continuing in High dose in the follow up period (8 months).
- Vehicle QID (4 Months) Plus .1% QID (8 Months Safety Follow-up): Participants in this group received Placebo in Period I (4 months) and continuing in High dose in the follow up period (8 months).
- Total High Dose; Total Low Dose: Total of participants that received High dose from the overall study period (0-12 months).
- .1% BID + Vehicle BID (4 Months) Plus .1% BID+ Vehicle BID (8 Months Safety Follow-up): Participants in this group received Low dose in Period I (4 months) and continuing in Low dose in the follow up period (8 months).
- Vehicle QID (4 Months) Plus .1% BID+ Vehicle BID (8 Months Safety Follow-up): Participants in this group received Placebo in Period I (4 months) and continuing in Low dose in the follow up period (8 months).
Arm/Group | .1% QID (4 Months) Plus .1% QID (8 Months Safety Follow-up) | Vehicle QID (4 Months) Plus .1% QID (8 Months Safety Follow-up) | Total High Dose | .1% BID + Vehicle BID (4 Months) Plus .1% BID+ Vehicle BID (8 Months Safety Follow-up) | Vehicle QID (4 Months) Plus .1% BID+ Vehicle BID (8 Months Safety Follow-up) | Total Low Dose
Serious Adverse Events (participants affected / at risk) | 3/50 | 0/22 | 3/72 | 1/44 | 0/26 | 1/70
Other Adverse Events (participants affected / at risk) | 29/50 | 13/22 | 42/72 | 24/44 | 11/26 | 35/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | .1% QID (4 Months) Plus .1% QID (8 Months Safety Follow-up) (N=50) | Vehicle QID (4 Months) Plus .1% QID (8 Months Safety Follow-up) (N=22) | Total High Dose (N=72) | .1% BID + Vehicle BID (4 Months) Plus .1% BID+ Vehicle BID (8 Months Safety Follow-up) (N=44) | Vehicle QID (4 Months) Plus .1% BID+ Vehicle BID (8 Months Safety Follow-up) (N=26) | Total Low Dose (N=70)
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | .1% QID (4 Months) Plus .1% QID (8 Months Safety Follow-up) (N=50) | Vehicle QID (4 Months) Plus .1% QID (8 Months Safety Follow-up) (N=22) | Total High Dose (N=72) | .1% BID + Vehicle BID (4 Months) Plus .1% BID+ Vehicle BID (8 Months Safety Follow-up) (N=44) | Vehicle QID (4 Months) Plus .1% BID+ Vehicle BID (8 Months Safety Follow-up) (N=26) | Total Low Dose (N=70)
Ocular hyperaemia (Eye disorders) | 2 | 2 | 4 | 0 | 1 | 1
Eye pruritus (Eye disorders) | 0 | 3 | 3 | 0 | 1 | 1
Corneal leukoma (Eye disorders) | 2 | 0 | 2 | 0 | 1 | 1
Ulcerative keratitis (Eye disorders) | 2 | 0 | 2 | 1 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 2
Foreign body sensation in eyes (Eye disorders) | 1 | 0 | 1 | 1 | 0 | 1
Ocular discomfort (Eye disorders) | 0 | 2 | 2 | 0 | 0 | 0
Abnormal sensation in eye (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Blepharitis (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Cataract subcapsular (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0
Conjunctival irritation (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Corneal deposits (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0
Corneal neovascularisation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Diplopia (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Eyelid erosion (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Meibomianitis (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 3 | 5 | 1 | 6
Influenza (Infections and infestations) | 4 | 0 | 4 | 0 | 0 | 0
Pharyngitis (Eye disorders) | 2 | 0 | 2 | 0 | 2 | 2
Tonsillitis (Infections and infestations) | 2 | 0 | 2 | 2 | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 2 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Conjunctivitis viral (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Eye infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Molluscum contagiosum (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Parasitic gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Instillation site pain (General disorders) | 6 | 4 | 10 | 5 | 0 | 5
Instillation site pruritus (General disorders) | 2 | 3 | 5 | 4 | 0 | 4
Instillation site erythema (General disorders) | 1 | 2 | 3 | 2 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 1 | 2 | 1 | 3
Application site discharge (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Application site erosion (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Application site swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Instillation site foreign body sensation (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Instillation site lacrimation (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 2
Allergic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 1 | 5 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Intraocular pressure decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Protein total increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Growing pains (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0 | 0
Removal of internal fixation (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes